CLINICAL TRIAL: NCT02434458
Title: Investigation of Sudoscan in the Evaluation of Small Fiber Dysfunction in Korean Patients With Autoimmune Disorders
Brief Title: Sudoscan in Patients With Autoimmune Disorders
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Assistant Professor, The Catholic University of Korea
Other Study IDs: HC15DISI0040
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Autoimmune Disease
Keywords: fibromyalgia,; polyneuropathy; small fiber neuropathy; rheumatoid arthritis; sudomotor
MeSH Terms: conditions — Autoimmune Diseases; Fibromyalgia; Polyneuropathies; Small Fiber Neuropathy; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Fibromyalgia case group: Patients diagnosed with fibromyalgia from the department of rheumatology will be subject to sudoscan evaluation and NCS studies.
- Control: Healthy control subjects
- Rheumatoid arthritis group: Patients diagnosed with rheumatoid arthritis at the department of rheumatology will be subject to sudoscan evaluation and NCS studies.

SUMMARY:
The purpose of this study is to assess the diagnostic utility of Sudoscan in assessing small fiber nerve function, specifically those of the sudomotor, in patients with autoimmune disorders (i.e fibromyalgia and rheumatoid arthritis).

DETAILED DESCRIPTION:
Small fiber neuropathy can manifest in different autonomic and painful symptoms, but current diagnostic tools are confined to nerve conduction studies and quantitative sensory testing.

The former can only asses the large nerve fibers and fail to reflect sudomotor function, the latter tool can be subject to technical error. Pain and autonomic dysfunction, which reflect small fiber dysfunction has recently gained much interest in disorders with polyneuropathy but current studies have been confined mostly to diabetic polyneuropathies. There has been growing evidence that autoimmune disorders such as fibromyalgia can also manifest in small fiber dysfunction. Because of the complexity of diagnosing small fiber dysfunction, there are yet no standard protocols on how to assess and treat these patients. Sudoscan uses reverse iontophoresis to assess the function of the sweat glands. The tool is easy to use, non-invasive with quantitative results that are objective.

The objective of this study is to assess the small fiber function; that is the sudomotor function; using Sudoscan in patients diagnosed with fibromyalgia and rheumatoid arthritis.

ELIGIBILITY:
Inclusion criteria:

A. for healthy control group

- No previous diagnosis of peripheral polyneuropathy, fibromyalgia or rheumatoid arthritis

B. For case group

* Fibromyalgia diagnosed by the rheumatology department
* Rheumatoid arthritis diagnosed by the the rheumatology department.

Exclusion Criteria:

For control group

-Participants with previously diagnosed with medical conditions that are known to cause peripheral polyneuropathy (i.e. diabetes mellitus, chronic renal failure, hepatitis, malnutrition), or participants taking medications related to peripheral polyneuropathy(chemoagents, anti Tbc medication) or manifest with symptoms and signs of tingling sensation and gait disturbance that indicate presence of underlying peripheral polyneuropathy.

For both control and case groups

* Severe skin deficits or swelling that may impede nerve conduction study
* Concomitant presence of mononeuropathy of the extremities.
* Past surgical or traumatic episodes of the foot and distal extremities subject to nerve conduction study
* History of chronic alcoholism, of history of heavy alcohol ingestion with the last 24 hours prior o exam
* Pregnant status at time of evaluation
* presence of pacemaker of defibrillator
* physical inability to lay the palms of the hand and soles of the feet on the plate electrodes.
* scars on the palm and soles of the feet that may impair recording from the plate electrodes
* venous insufficiency, foot swelling or foot ulceration or infection
* Abnormal fasting glucose or Vit B12, thyroid dysfunction, Vit D and abnormal levels of lipid profile, HbA1c > 7
* Medications with anticholinergics, TCA, anti-histamine, anti-muscarinic medication within the last 48hours
* Patients currently taking Anti Parkinson agents, ranitidine, or other muscle relaxants, beta blockers and atropine
* Heavy alcohol ingestion within the last 24 hour

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who meet the following diagnostic criteria for either 1. Fibromyalgia or 2. Rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sudoscan values | once at time of enrollment
  Small fiber function from sweat glands, using Sudoscan

SECONDARY OUTCOMES:
NCS studies | once at time of enrollment
  NCS values of the upper and lower extremity sensory nerves performed by an electromyographer

CONTACTS AND LOCATIONS:
Overall Officials: Su-Jin Monn, M.D., PhD, Study Director — Catholic University of Korea, College of Medicine Bucheon St. Mary's Hospital
Locations (2):
- South Korea (2):
  - Bucheon St Mary's Hospital, Catholic University of Korea, Bucheon-si, Gyenoggido
  - Bucheon St Mary's Hospital, Bucheon-si